CLINICAL TRIAL: NCT00193453
Title: A Phase II Trial of First-Line Therapy With Gemcitabine, Docetaxel, and Cetuximab in Patients With Unresectable Stage III or IV Non-Small Cell Lung Cancer
Brief Title: Gemcitabine, Docetaxel, and Cetuximab in Patients With Unresectable Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 92
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2012-11-13 (Estimated); Last update posted 2012-11-13 (Estimated); Status verified 2012-10

CONDITIONS: Lung Cancer
Keywords: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Gemcitabine; Docetaxel; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Newly-diagnosed unresectable stage III/IV NSCLC patients were treated with docetaxel-30mg/m2 IV; gemcitabine-1000mg/m2 IV days 1, 8; cetuximab-400mg/m2 IV day 1, then 250 mg/m2 IV weekly. Patients received up to 6 cycles (21-d).
  Interventions: Drug: Gemcitabine; Drug: Docetaxel; Drug: Cetuximab

INTERVENTIONS:
Drug: Gemcitabine — 1000mg/m2 30min IV, Day 1 & 8
  Other Names: Gemzar
Drug: Docetaxel — 30mg/m2, 30min IV, day 1 & 8
  Other Names: Taxotere
Drug: Cetuximab — 100mg/m2 IV, Cycle 1 Day 1, 250mg/m2 IV day 8 & 15, all subsequent cycles 250mg/m2 IV day 1, 8, & 15
  Other Names: Erbitux

SUMMARY:
This purpose of this study is to evaluate the role of gemcitabine and docetaxel, a well tolerated chemotherapy regimen in the treatment of advanced non-small cell lung cancer (NSCLC), in combination with a novel agent cetuximab.

DETAILED DESCRIPTION:
Upon determination of eligibility all patients will receive:

* Docetaxel + Gemcitabine + Cetuximab

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, you must meet the following criteria:

* 18 years of age or older
* Non-small cell lung cancer confirmed by biopsy
* Unresectable stage III or IV disease
* Measurable disease
* Must not have received any prior chemotherapy for lung cancer
* Able to perform activities of daily living without considerable assistance
* Adequate bone marrow, kidney, and liver function
* Signed informed consent

Exclusion Criteria:

You cannot participate in the study if any of the following apply to you:

* History of serious heart disease within six months prior to study entry
* Prior treatment with agents that target the EGFR pathway
* History of any other uncontrolled or significant disease

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have. You can then decide if you wish to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-07; Primary Completion 2009-02 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Spigel, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (10):
- United States (10):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Northeast Arkansas Clinic, Jonesboro, Arkansas
  - Florida Cancer Specialists, Fort Myers, Florida
  - Gainsville Hematology Oncology Associates, Gainesville, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Graves-Gilbert Clinic, Bowling Green, Kentucky
  - Consultants in Blood Disorders and Cancer, Louisville, Kentucky
  - Mercy Hospital, Portland, Maine
  - Consultants in Medical Oncology and Hematology, Drexel Hill, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- [Result] Spigel DR, Greco FA, Thompson DS, Webb C, Rubinsak J, Inhorn RC, Reeves J Jr, Vazquez ER, Lane CM, Burris HA 3rd, Hainsworth JD. Phase II study of cetuximab, docetaxel, and gemcitabine in patients with previously untreated advanced non-small-cell lung cancer. Clin Lung Cancer. 2010 May;11(3):198-203. doi: 10.3816/CLC.2010.n.026. PMID 20439197
- See also: Published article in Clinical Lung Cancer — http://cigjournals.metapress.com/content/wt0106p0206m0q67/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention
Started | 69
Completed | 21
Not Completed | 48

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 51
Age Continuous [Mean (Standard Deviation); unit: years] | 68 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 48
Region of Enrollment [Number; unit: participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Overall Clinical Response Rate
Description: Overall response rate was defined as the proportion of treated patients whose best response was a complete or partial response after completing at least two courses of treatment.
Time Frame: 18 months
Population: Patients with at least one restaging were assessed for overall clinical response. Patients who died prior to the first restaging or were not assessed due to physician/patient discretion were not included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Intervention
Number analyzed (Participants) | 65
Percentage of participants | 17 [9 to 29]

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival was defined as the interval between the start date of treatment and the date of occurrence of progressive disase or death from any cause.
Time Frame: 18 months
Population: All patients were assessed for progression-free survival.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intervention
Number analyzed (Participants) | 69
Months | 4.0 [2.7 to 5.9]

3. Secondary Outcome: Response Duration
Description: The Response Duration was calculated from time of initial measured response to date of first observation of progressive disease.
Time Frame: 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Intervention
Number analyzed (Participants) | 65
Months | 7.0 [2.5 to 8.9]

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 43/69
Other Adverse Events (participants affected / at risk) | 69/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=69)
Acute Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Allergic reaction (Immune system disorders) | 3
Atrial fibrillation (Cardiac disorders) | 4
Cardiac Arrhythmia - Other (Abnormal EKG) (Cardiac disorders) | 1
Cardiac Arrythmia (NOS) (Cardiac disorders) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 4
Cardiopulmonary arrest (Cardiac disorders) | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 2
Death not associated with CTCAE term - Disease Progression NOS (General disorders) | 6
Dehydration (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Edema (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 2
Fever (General disorders) | 1
Hemorrhage, GI - Peritoneal cavity (Blood and lymphatic system disorders) | 1
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 1
Infection - Other (Cellulitis) (Infections and infestations) | 1
Infection - Other (Pneumonia) (Infections and infestations) | 5
Neutrophils (Blood and lymphatic system disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other (Respiratory Arrest) (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other (Hypoxic respiratory failure) (Respiratory, thoracic and mediastinal disorders) | 1
Renal failure (Renal and urinary disorders) | 2
Supraventricular arrhythmia NOS (Cardiac disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 5
Vascular - Other (Bilateral carotid occlusion) (Vascular disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=69)
Alopecia (Skin and subcutaneous tissue disorders) | 15
Hemoglobin (Blood and lymphatic system disorders) | 46
Anorexia (Gastrointestinal disorders) | 30
Pain - joints (Musculoskeletal and connective tissue disorders) | 13
Cardiac Toxicities (Infarction, Arrythmia) (Cardiac disorders) | 19
Constipation (Gastrointestinal disorders) | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dehydration (Gastrointestinal disorders) | 5
Diarrhea (Gastrointestinal disorders) | 34
Dizziness (Nervous system disorders) | 4
Taste Alteration (Gastrointestinal disorders) | 8
Edema (Blood and lymphatic system disorders) | 26
Hemorrhage, pulmonary/upper respiratory - Nose (Blood and lymphatic system disorders) | 5
Fatigue (General disorders) | 56
Fever (NOS) (General disorders) | 11
Hyperglycemia (Metabolism and nutrition disorders) | 10
Watery eye (Eye disorders) | 4
Allergic Reaction (Immune system disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 25
Hyponatremia (Metabolism and nutrition disorders) | 4
Hypotension (Cardiac disorders) | 4
Infection (NOS) (Infections and infestations) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 4
Leukocytes (Blood and lymphatic system disorders) | 6
Mucositis (Gastrointestinal disorders) | 19
Pain - muscles (Musculoskeletal and connective tissue disorders) | 11
Nail changes (Skin and subcutaneous tissue disorders) | 8
Nausea (Gastrointestinal disorders) | 31
Neutrophils (Blood and lymphatic system disorders) | 30
Pain (NOS) (General disorders) | 41
Pulmonary Toxicities (dyspnea, pulmonary embolism) (Respiratory, thoracic and mediastinal disorders) | 43
Neuropathy-sensory (Nervous system disorders) | 9
Skin toxicities (Skin and subcutaneous tissue disorders) | 59
Platelets (Blood and lymphatic system disorders) | 39
Vomiting (Gastrointestinal disorders) | 14
Flu-like syndrome (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.